CLINICAL TRIAL: NCT07147062
Title: Comparison of the Postoperative Analgesic Effects of Rectus Sheath Block and Caudal Epidural Block in Pediatric Patients Scheduled for Percutaneous Internal Ring Suturing
Brief Title: Comparison of the Postoperative Analgesic Effects of RSB and CEB in Pediatric Patients Scheduled for Percutaneous Internal Ring Suturing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-170
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Percutaneous Internal Ring Suturing; Pain Management
Keywords: Percutaneous internal ring suturing; Rectus sheath block; Caudal epidural block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus Sheath Block (Active Comparator): Using an in-plane approach from cephalad to caudal, a 22G, 50-mm needle will be advanced through the subcutaneous tissues, penetrating the anterior rectus sheath and progressing within the muscle until the needle tip contacts the posterior rectus sheath. After negative aspiration, a total volume of 0.5 mL/kg of 0.25% bupivacaine-distributed equally between both sides-will be injected bilaterally under direct ultrasound guidance.
  Paracetamol at a dose of 10 mg/kg will be administered intraoperatively.
  Interventions: Procedure: Rectus Sheath Block
- Caudal Epidural Block (Active Comparator): A 22G caudal epidural needle will be inserted at approximately a 45° angle toward the sacral hiatus, and the characteristic "click" sensation will be felt upon passing the sacrococcygeal ligament. The needle will then be advanced carefully in the cephalad direction, parallel to the longitudinal axis of the spinal canal. After confirming correct placement by negative aspiration, 1 mL/kg of 0.25% bupivacaine will be administered.
  Paracetamol at a dose of 10 mg/kg will be administered intraoperatively.
  Interventions: Procedure: Caudal Epidural Block

INTERVENTIONS:
Procedure: Rectus Sheath Block — A total volume of 0.5 mL/kg of 0.25% bupivacaine-distributed equally between both sides-will be injected bilaterally under direct ultrasound guidance.
  Arms: Rectus Sheath Block
Procedure: Caudal Epidural Block — A 22G caudal epidural needle will be inserted at approximately a 45° angle toward the sacral hiatus, and the characteristic "click" sensation will be felt upon passing the sacrococcygeal ligament. The needle will then be advanced carefully in the cephalad direction, parallel to the longitudinal axis of the spinal canal. After confirming correct placement by negative aspiration, 1 mL/kg of 0.25% bupivacaine will be administered.
  Arms: Caudal Epidural Block

SUMMARY:
Inguinal hernia is one of the most common surgical pathologies in children, and the minimally invasive percutaneous internal ring suturing (PIRS) technique is widely preferred.

By providing effective pain control, nerve blocks reduce postoperative opioid requirements, thereby minimising opioid-related adverse effects and lowering the risk of pulmonary and cardiovascular complications.

This study aims to compare the postoperative analgesic effects of rectus sheath block and caudal epidural block in pediatric patients undergoing PIRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 1 and 8 years
* ASA physical status I-II
* Patients who underwent PIRS surgery in the operating room and received either a rectus sheath block or a caudal epidural block

Exclusion Criteria:

* Patients younger than 1 year or older than 8 years
* ASA physical status ≥ III
* History of bleeding diathesis

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | On the operation day
  Pain will be assessed at rest and during coughing using the FLACC (Face, Legs, Activity, Cry, Consolability) scale, scored from 0 to 10. Pain assessments will be performed at the 0th, 1st, 2nd, 4th, 12th, and 24th hours after surgery.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | On the operation day
  The occurrence of postoperative nausea and vomiting (PONV) and the number of episodes will be recorded.
Time to first mobilization | On the operation day
  Time to first mobilization will be recorded in hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)